CLINICAL TRIAL: NCT04228965
Title: A Prospective Trial of Varenicline and Incentives for Tobacco Cessation in Adults
Brief Title: Cannabis and Tobacco Co-use Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Erin McClure, Principal Investigator, Medical University of South Carolina
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00086954; R37CA237245 (NIH)
Record Dates: First submitted 2019-12-11; First posted 2020-01-14 (Actual); Results first posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Tobacco Use Disorder
Keywords: Smoking Cessation
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Varenicline; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Co-Use Group (Other): Cannabis and tobacco co-use group.
  Interventions: Drug: Varenicline; Behavioral: Contingency Management; Behavioral: Counseling
- Tobacco Only Group (Active Comparator): Tobacco only group.
  Interventions: Drug: Varenicline; Behavioral: Contingency Management; Behavioral: Counseling

INTERVENTIONS:
Drug: Varenicline — Varenicline is a medication approved by the Food and Drug Administration for the treatment of tobacco use disorder among adults (ages 18 and over). In this study, all participants will be administered active medication for the recommended 12 week treatment period. The standard dose titration schedule will be used, which includes 0.5 mg once per day (q.d.) on Days 1-3, 0.5 mg twice per day (b.i.d.) on Days 4-7, and 1.0 mg b.i.d. starting on Day 8. Dosing of 2.0 mg per day will be maintained for the next 11 weeks, for a total of 12 weeks of active treatment for all study participants.
  Other Names: Chantix
Behavioral: Contingency Management — Contingency management procedures will be implemented and financial incentives will be provided at weekly visits contingent on tobacco abstinence verified through urinary qualitative cotinine (starting at Week 2). A set amount of $20 per study visit will be delivered based on a negative qualitative urinary cotinine result.
Behavioral: Counseling — Psychosocial counseling will be administered by trained research staff leading up to the target quit date and throughout the study. Counseling will include motivational enhancement for medication adherence and tobacco cessation. The content of counseling will be skills-based and will focus on enlisting social support, recognizing smoking triggers, managing craving/withdrawal/stress, etc.

SUMMARY:
The purpose of this study is to better understand tobacco outcomes using a well-known stop smoking medication, varenicline, and financial incentives with tobacco users. The investigators are also interested in how cannabis/marijuana and tobacco interact during a tobacco quit attempt. All participants will receive tobacco cessation treatment (varenicline) for 12 weeks. This study will recruit adult tobacco users (ages 18-40) who are motivated to quit smoking cigarettes.

DETAILED DESCRIPTION:
Cannabis co-use among tobacco users is exceedingly common and rates of co-use appear to be increasing among adults in the US, which is consistent with overall increases in cannabis use rates among US adults. Given the current cannabis landscape, further increases in cannabis use are likely and may result in continued increases in the co-use of cannabis and tobacco.

Despite high rates of co-use, there is little consensus regarding treatment recommendations for this population and an understanding of the impact of co-use on successful cessation. The literature on the impact of co-use on tobacco cessation outcomes specifically has been mixed and fraught with limitations, including methodological variation, lack of biochemical verification to confirm cannabis use status and severity, and variations in study samples. Currently, no prospective studies have been conducted to evaluate the impact of cannabis use on tobacco cessation outcomes. Further, no studies have collected cannabis use changes during tobacco cessation treatment to assess for concurrent reductions, abstinence, or of greater concern, compensatory (i.e., increased) use as a result of tobacco reduction/abstinence.

This study is a prospective 12-week tobacco cessation trial using established methods and outcomes typical of tobacco cessation trials, but specifically recruiting co-users of cannabis. The aims of this proposed study are to; 1) examine the impact of cannabis co-use on tobacco cessation outcomes among co-users compared to tobacco only participants (Aim #1), 2) among cannabis co-users, assess changes in cannabis use during tobacco treatment (Aim #2), and 3) assess for a dose-dependent impact of cannabis co-use severity on tobacco cessation (Exploratory Aim #1).

ELIGIBILITY:
Inclusion Criteria:

1. Between the ages of 18 and 40 years old
2. Must be able to understand the study and provide written informed consent
3. Daily cigarette smoker for ≥ 6 months, smoking ≥ 5 cigarettes per day
4. Must submit a breath carbon monoxide (CO) sample of ≥ 7 parts per million (ppm) at the screening visit
5. Be interested in quitting smoking tobacco cigarettes (defined as a 5 or above on a 10-point Likert scale assessing interest in quitting [1=not at all interested, 10=extremely interested])
6. Must be willing to take varenicline for the standard 12-week course of treatment
7. If female, agreement to use birth control (any form) to avoid pregnancy during study procedures

   Additional inclusion criteria will be implemented for cannabis co-users, which include:
8. Self-reported use of cannabis on at least 10 out of the past 30 days or submit a positive qualitative urinary cannabinoid test at screening (limit of detection is 50 ng/ml)

Exclusion Criteria:

1. Any serious or unstable medical/psychiatric disorder (including severe substance use disorders, other than cannabis or tobacco use disorders) or other significant concern in the past three months that may interfere with study performance, impact participant safety, compliance with study procedures, or potentially confound the interpretation of findings
2. Currently pregnant, lactating, or contemplating pregnancy in the next 6 months
3. Current use of medications with smoking cessation efficacy
4. Use of any medications that would interfere with varenicline
5. No regular use of other tobacco or nicotine products other than combustible cigarettes (e.g., smokeless tobacco, electronic cigarettes, etc.) in the past month prior to the quit attempt

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin McClure, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (3):
- United States (3):
  - Medical University of South Carolina - Charleston, Charleston, South Carolina
  - Medical University of South Carolina - Florence, Florence, South Carolina
  - Behavioral Health Services of Pickens County, Pickens, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walters KJ, Baker NL, Tomko RL, Gray KM, Carpenter MJ, McClure EA. Determining the impact of cannabis use and severity on tobacco cessation outcomes: study protocol for a prospective tobacco treatment trial. BMC Psychol. 2023 Jan 25;11(1):25. doi: 10.1186/s40359-023-01060-2. PMID 36698194

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the community at three sites across South Carolina, USA; MUSC Charleston (Charleston, SC), Behavioral Health Services of Pickens County (BHS, Pickens, SC) and MUSC Florence (Florence, SC). Enrollment ran from January 2020 until March 2024, with the MUSC Florence site being added in 2022. A total of 259 participants were screened for eligibility and 181 (70%) were enrolled
Period: Overall Study
Arm/Group | Co-Use Group | Tobacco Only Group
Started | 110 | 71
Completed | 66 | 55
Not Completed | 44 | 16
Not completed — Lost to Follow-up | 26 | 11
Not completed — Withdrawal by Subject | 18 | 5

BASELINE CHARACTERISTICS:
Population: A total of 181 participants were enrolled (dispensed study medication): 110 in the cannabis co-use cohort and 71 in the tobacco-only cohort.
Groups:
- Total: Total of all reporting groups
Arm/Group | Co-Use Group | Tobacco Only Group | Total
Number analyzed (Participants) | 110 | 71 | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.3 (5.6) | 34.5 (5.1) | 33.1 (5.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender Identity: Woman | 47 | 42 | 89
  Gender Identity: Man | 62 | 27 | 89
  Gender Identity: Other/Unknown | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 42 | 89
  Male | 63 | 29 | 92
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 3 | 11
  Not Hispanic or Latino | 102 | 68 | 170
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 29 | 5 | 34
  White | 73 | 62 | 135
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 110 | 71 | 181
Cigarettes per day (assessed in the 30 days prior to screening/baseline)) [Mean (Standard Deviation); unit: cigarettes per day] | 13.4 (7.8) | 14.9 (7.2) | 14.1 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Biologically Verified 7-day Point Prevalence Tobacco Abstinence at the End of Treatment (Week 12)
Description: 7-day point prevalence abstinence from tobacco at the end of treatment (Week 12) will be assessed via biochemical verification (urinary cotinine; ng/ml) and will be compared between cannabis co-users and tobacco only controls.
Time Frame: Final 7 days of treatment (Week 12)
Population: Estimation of the primary outcome was completed using 3 methods: 1) simple imputation (missing=smoking), 2) methods of multiple imputation, and 3) utilizing all available data (number analyzed is lower in each compared to imputation methods).
Measure: Count of Participants; unit: Participants
Groups:
- Co-Use Group: Cannabis and tobacco co-use group, defined as use of cannabis on 10+ out of the past 30 days or submitted a positive qualitative urinary cannabinoid test at screening.
  Varenicline: Varenicline is a medication approved by the Food and Drug Administration for the treatment of tobacco use disorder among adults (ages 18 and over). In this study, all participants will be administered active medication for the recommended 12 week treatment period. The standard dose titration schedule will be used, which includes 0.5 mg once per day (q.d.) on Days 1-3, 0.5 mg twice per day (b.i.d.) on Days 4-7, and 1.0 mg b.i.d. starting on Day 8. Dosing of 2.0 mg per day will be maintained for the next 11 weeks, for a total of 12 weeks of active treatment for all study participants.
  Contingency Management: Financial incentives will be provided at weekly visits contingent on tobacco abstinence verified through urinary qualitative cotinine (starting at Week 2). A set amount of $20 per study visit will be delivered based on a negative qualitative urinary cotinine result.
  Counseling: Psychosocial counseling will be administered by trained research staff leading up to the target quit date and throughout the study. Counseling will include motivational enhancement for medication adherence and tobacco cessation. The content of counseling will be skills-based and will focus on enlisting social support, recognizing smoking triggers, managing craving/withdrawal/stress, etc.
- Tobacco Only Group: Tobacco only group, defined as ≥ 5 cigarettes per day and not using cannabis 10 or more days in the past 30 nor submitting a positive qualitative urinary cannabinoid test at screening.
  Varenicline: Varenicline is a medication approved by the Food and Drug Administration for the treatment of tobacco use disorder among adults (ages 18 and over). In this study, all participants will be administered active medication for the recommended 12 week treatment period. The standard dose titration schedule will be used, which includes 0.5 mg once per day (q.d.) on Days 1-3, 0.5 mg twice per day (b.i.d.) on Days 4-7, and 1.0 mg b.i.d. starting on Day 8. Dosing of 2.0 mg per day will be maintained for the next 11 weeks, for a total of 12 weeks of active treatment for all study participants.
  Contingency Management: Financial incentives will be provided at weekly visits contingent on tobacco abstinence verified through urinary qualitative cotinine (starting at Week 2). A set amount of $20 per study visit will be delivered based on a negative qualitative urinary cotinine result.
  Counseling: Psychosocial counseling will be administered by trained research staff leading up to the target quit date and throughout the study. Counseling will include motivational enhancement for medication adherence and tobacco cessation. The content of counseling will be skills-based and will focus on enlisting social support, recognizing smoking triggers, managing craving/withdrawal/stress, etc.
Arm/Group | Co-Use Group | Tobacco Only Group
Number analyzed (Participants) | 110 | 71
Participants
  Number of Participants with 7-day Point Prevalence Abstinence: Simple Imputation | 30 | 40
  Number of Participants with 7-day Point Prevalence Abstinence: Multiple Imputation | 36 | 42
  Number of Participants with 7-day Point Prevalence Abstinence: Available Data: number analyzed (Participants) | 74 | 62
  Number of Participants with 7-day Point Prevalence Abstinence: Available Data | 30 | 40

2. Secondary Outcome: Cannabis Use During Tobacco Cessation Treatment (Among Co-users)
Description: Among cannabis co-users (n=110), cannabis use (based on urinary cannabinoids [ng/ml]) during the final 4 weeks of tobacco treatment (Weeks 9-12) will be assessed.
Time Frame: Final 4 weeks of study treatment (Weeks 9-12)
Population: All participants in the cannabis co-use group (n=110) with any data available during the final 4 weeks of study treatment (weeks 9-12). A total of 75 participants had data available for at least one of the final 4 weekly visits. The tobacco-only group was not included in this outcome.
Measure: Geometric Mean (Standard Error); unit: urinary cannabinoids in ng/ml
Arm/Group | Co-Use Group | Tobacco Only Group
Number analyzed (Participants) | 75 | 0
urinary cannabinoids in ng/ml
  Week 9 urinary cannabinoids [ng/ml]: number analyzed (Participants) | 59 | 0
  Week 9 urinary cannabinoids [ng/ml] | 405 (96) |
  Week 10 urinary cannabinoids [ng/ml]: number analyzed (Participants) | 60 | 0
  Week 10 urinary cannabinoids [ng/ml] | 402 (98) |
  Week 11 urinary cannabinoids [ng/ml]: number analyzed (Participants) | 60 | 0
  Week 11 urinary cannabinoids [ng/ml] | 376 (86) |
  Week 12 urinary cannabinoids [ng/ml]: number analyzed (Participants) | 73 | 0
  Week 12 urinary cannabinoids [ng/ml] | 414 (88) |

ADVERSE EVENTS:
Time Frame: Adverse events were collected starting after study screening and up to 6 months following the screening assessment and through the Week 26 follow-up study visit.
Description: Other non-serious adverse events that occured in greater than 5% of participants (in either experimental group) are reported here. Each adverse event was coded with a MedDRA term and the specific Adverse Event term is used.
Arm/Group | Co-Use Group | Tobacco Only Group
All-Cause Mortality (participants affected / at risk) | 0/110 | 0/71
Serious Adverse Events (participants affected / at risk) | 1/110 | 1/71
Other Adverse Events (participants affected / at risk) | 76/110 | 56/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Use Group (N=110) | Tobacco Only Group (N=71)
Gastrointestinal Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Altered State of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-Use Group (N=110) | Tobacco Only Group (N=71)
Vomiting (Gastrointestinal disorders) | 6 (6) | 1 (1)
Nausea (Gastrointestinal disorders) | 31 (40) | 22 (27)
Irritability (General disorders) | 10 (11) | 3 (3)
Weight gain (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 7 (8) | 6 (6)
Somnolence (Nervous system disorders) | 4 (4) | 4 (4)
Vivid Dreams (Psychiatric disorders) | 22 (24) | 23 (29)
Depressed mood (Psychiatric disorders) | 6 (7) | 3 (3)
Insomnia (Psychiatric disorders) | 6 (6) | 5 (7)
Anxiety (Worsening) (Psychiatric disorders) | 6 (6) | 2 (5)
Tobacco Withdrawal Symptoms (Psychiatric disorders) | 2 (2) | 4 (4)
Vivid Dreams (Worsening) (Psychiatric disorders) | 5 (7) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/65/NCT04228965/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-06): https://cdn.clinicaltrials.gov/large-docs/65/NCT04228965/ICF_000.pdf